CLINICAL TRIAL: NCT04073784
Title: An Open-Label, Single Center, Nonrandomized, Phase 1 Study to Evaluate Safety and Efficacy of Gemcitabine Combined With Apatinib and Toripalimab in Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Gemcitabine Combined With Apatinib and Toripalimab in Recurrent or Metastatic Nasopharyngeal Carcinoma.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-BYK-GAT2019
Record Dates: First submitted 2019-08-25; First posted 2019-08-29 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Toripalimab; Gemcitabine; Apatinib; recurrent NPC; metastatic NPC
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: Subjects receive Apatinib for oral administration, 250mg, once a day, gemcitabine 1000mg/m2 (Day 1 and Day 8) and Toripalimab , 240mg, (Day 1) of each 21days for at most 6 cycles, followed by Toripalimab 240mg every three weeks (Q3W) and Apatinib 250mg once a day maintenance for the remainder of the study or until documented PD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitabine combined with Apatinib and Toripalimab (Experimental): Subjects receive Apatinib for oral administration, 250mg, once a day, gemcitabine 1000mg/m2 (Day 1 and Day 8) and Toripalimab , 240mg, (Day 1) of each 21days for at most 6 cycles, followed by Toripalimab 240mg every three weeks (Q3W) and Apatinib 250mg once a day maintenance for the remainder of the study or until documented PD.
  Interventions: Drug: Gemcitabine combined with Aptinib and Toripalimab

INTERVENTIONS:
Drug: Gemcitabine combined with Aptinib and Toripalimab — Gemcitabine injection, gemcitabine 1000mg/m2, Day 1 and Day 8 of each 21 day, maximum 6 cycles.
  Apatinib for oral administration, 250mg, once a day. Apatinib maintenance.
  Toripalimab injection, 240mg, Day 1 each 21day. Toripalimab maintenance.

SUMMARY:
This is an open-label, single center, non-randomized, phase I trial to evaluate the safety and efficacy of gemcitabine combined with apatinib and toripalimab in patients with the recurrent or metastatic nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This is an open-label, single center, non-randomized, phase I trial to evaluate the safety and efficacy of gemcitabine combined with apatinib and toripalimab in patients with the recurrent or metastatic nasopharyngeal carcinoma.

Safety evaluations (both clinical and laboratory) are performed at baseline, before each study treatment, and throughout the study.Tumor response will be assessed by radiographic examination in screening visit and every 2 cycles after first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-70 years of age.
2. Subjects diagnosed with pathological confirmed Primary metastatic nasopharyngeal carcinoma, or subjects with recurrent NPC that is unfit for local treatment.
3. Subjects with recurrent and metastatic NPC who did't receive any Systemic chemotherapy, neoadjuvant chemotherapy, concurrent radiochemotherapy and adjuvant chemotherapy 6 month before first dose are excepted.
4. ECOG performance status of 0 or 1.
5. Life expectancy more than 12 weeks.
6. Subjects enrolled must have measurable lesion(s) according to response evaluation criteria in solid (RECIST) v1.1.
7. Adequate organ function assessed by laboratory parameters during the screening period
8. Female subjects agree not to be pregnant or lactating from beginning of the study screening through at least 3 months after receiving the last dose of study treatment. Both men and women of reproductive potential must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy. A highly effective method of contraception is defined as one that results in a low failure rate, that is, less than 1% per year when used consistently and correctly
9. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Subjects with any active autoimmune disease or history of autoimmune disease, or history of syndrome that requires systemic steroids or immunosuppressive medications, including but not limited to the following: rheumatoid arthritis, pneumonitis, colitis (inflammatory bowel disease), hepatitis, hypophysitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Subjects with the following conditions will not be excluded from this study: asthma that requires intermittent use of bronchodilators, hypothyroidism stable on hormone replacement, vitiligo, Graves' disease, or Hashimoto's disease. Additional exceptions may be made with medical monitor approval;
2. Known history of hypersensitivity to any components of the Toripalimab formulation;
3. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration. Note: corticosteroids used for the purpose of IV contrast allergy prophylaxis are allowed;
4. Active central nervous system (CNS) metastases (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive disease);
5. Uncontrolled clinically significant medical condition, including but not limited to the following:

   1. congestive heart failure (New York Health Authority Class > 2),
   2. unstable angina,
   3. myocardial infarction within the past 12 months,
   4. clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
6. Active infection or an unexplained fever; 38.5℃ during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, subjects with tumor fever may be enrolled);
7. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease;
8. Any other medical (eg, pulmonary, metabolic, congenital, endocrinal, or CNS disease), psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results;
9. Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation based on institutional guidelines and tests. Testing may include the following: HBV DNA, HCV RNA, hepatitis B surface antigen, or anti-Hepatitis B core antibody.
10. Subjects with hypertension (even with antihypertensive treatment) unable to reduce to the normal range. (Systolic blood pressure >140 mmHg/diastolic blood pressure > 90 mmHg ). Coronary heart disease, arrhythmia ≥II (including QTc lengthened, men > 450 ms, women > 470 ms) and cardiac failure.
11. Coagulation abnormalities (PT>16s、APTT>43s、TT>21s、Fbg<2g/L), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
12. Patients with or previous with serious hemorrhage (bleeding > 30 ml within 3 months), haemoptysis (> 5 ml within 4 weeks) of thromboembolic events within 12 months (including stroke events and/or transient ischemic attack).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-06-08 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 12months
  The safety will be assessed by ongoing reviews of clinical laboratory tests, Eastern Cooperative Oncology Group (ECOG) performance status, physical examination, electrocardiogram (ECG), and adverse events. Evaluations of immune safety will also be conducted (immune-related adverse events (AEs), or labs of autoimmune sera, inflammatory events, and immunogenicity). Safety evaluations (both clinical and laboratory) are performed at baseline, before each study treatment, and throughout the study.

SECONDARY OUTCOMES:
The proportion of patients who achieved an objective response | 12 months
  Defined as those with radiologically confirmed complete or partial response according to RECIST 1.1 assessed by the investigator;
The proportion of patients who achieved disease control, | 12months
  Defined as those with RECIST-defined objective response or stable disease;
The proportion of patients who achieved clinical benefit | 12 months
  Defined as those with confirmed objective response or stable disease that lasted for at least 6 months;
Progression-free survival (median and at 6 and 12 months) | 12 months
  Defined from the enrolment to RECISTdefined progression or death from any causes;
Duration of response | 12 months
  Defined as the time from first documentation of objective response to radiological disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] You R, Zou X, Ding X, Zhang WJ, Zhang MX, Wang X, Xu HS, Liu YL, Ouyang YF, Duan CY, Gu CM, Wang ZQ, Liu YP, Hua YJ, Huang PY, Chen MY. Gemcitabine combined with apatinib and toripalimab in recurrent or metastatic nasopharyngeal carcinoma. Med. 2022 Oct 14;3(10):664-681.e6. doi: 10.1016/j.medj.2022.07.009. Epub 2022 Aug 29. PMID 36041429